CLINICAL TRIAL: NCT06065189
Title: Evaluation and Promotion of Key Technologies of Base-edited Autologous Hematopoietic Stem Cell Transplantation in Treating Patients With β-thalassemia Major
Brief Title: Base-edited Autologous Hematopoietic Stem Cell Transplantation in Treating Patients With β-thalassemia Major
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: CorrectSequence Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-101-03
Record Dates: First submitted 2023-09-27; First posted 2023-10-03 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CS-101 injection (Experimental): Autologous CD34+(cluster of differentiation 34) hematopoietic stem cell suspension modified by in vitro base editing technique
  Interventions: Biological: CS-101 injection

INTERVENTIONS:
Biological: CS-101 injection — Autologous CD34+ hematopoietic stem cell suspension modified by in vitro base editing technique

SUMMARY:
The goal of this open label, single-arm clinical study is to learn about the safety and efficacy of base-edited autologous hematopoietic stem cell transplantation(CS-101) in treating patients with β-thalassemia major.

DETAILED DESCRIPTION:
CS-101 is an autologous CD34+ cell suspension modified by ex vivo base editing technology, removing the inhibitory effect of BCL11A on the γ-globin coding gene, inducing the production of γ-globin chains, increasing the concentration of fetal hemoglobin (HbF) in the blood, compensating for the loss of adult hemoglobin (HbA) to treat transfusion-dependent type/ Major β - thalassemia. The therapy addresses two major challenges in the treatment of the disease: lack of matching donors and graft-versus-host responses commonly seen in allogeneic hematopoietic stem cell transplantation.

The study consists of the following five phases:

Screening phase: Sign informed consent, complete screening assessments, and confirm the eligibility for enrollment; Baseline: check the subject's baseline status; Mobilization, collection and manufacturing phase: mobilize, collect autologous CD34+ cells and manufacture, release and transport CS-101 product; Conditioning and treatment phase: including myeloablation and CS-101 product infusion; Follow-up phase: 180 days post-infusion.

ELIGIBILITY:
Inclusion Criteria:

* 3 to 17 years old(inclusive) male or female subjects at the time of informed consenting
* Diagnosis of β-thalassemia, genotypes include but are not limited to β+β0, βEβ0, β0β0, etc
* Generally in good condition, Karnofsky performance score≥60 points for subjects≥16 years old at the time of autologous hematopoietic stem cell collection, or Lansky Play-Performance score≥60 points for subjects under 16 years old, or equivalent clinical evaluation as the investigator site's common practice
* For female subjects of childbearing potential: use effective contraceptive measures for at least 1 month prior to screening and agree to continue using such measures for contraception throughout the study
* For male subjects who have a potential ability to father a child: use condoms or other methods continuously from the start of mobilization to ensure effective contraception for sexual partners during the study period

Exclusion Criteria:

* Treatment with other investigational medications or other experimental interventions 30 days prior to signing informed consent or within 6 half-lives of the drug, whichever is longer.
* Subjects who have received or are receiving thalidomide and/or Luspatercept, when their drug-drug interaction on the efficacy and safety of CS-101 cannot be ruled out, unless at least there are 3 test results showing the total hemoglobin level before transfusion is below 9g/dL in the past 6 months before screening.
* Previously received allogeneic hematopoietic stem cell transplantation or gene(edited) therapy.
* Subjects have available related fully matching donors and are eligible and prepared for allogeneic hematopoietic stem cell transplantation.
* Subjects with coexisting α-thalassemia and more than 2 deletions or non-deletional mutations in the α-globin chain coding genes.
* Known to be allergic to drugs used during autologous hematopoietic stem cell transplantation (including but not limited to granulocyte colony-stimulating factor, busulfan, dextran), excipients(such as dimethyl sulfoxide), or instruments(such as intravenous catheters) as determined by the investigator are deemed unsuitable to participate in this study.
* Those with active infections, including but not limited to: HIV, hepatitis B, hepatitis C, cytomegalovirus, Epstein-Barr virus and treponema pallidum test positive, or known tuberculosis, parasitic infection, etc. who are judged by the investigator to be unsuitable to participate in this study
* Echocardiography results with ejection fraction below 45%
* Subjects who are febrile (temperature over 37.3° C) should be held back from enrolment.
* Advanced liver disease, defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT) >3 × upper limit of normal (ULN) or baseline International Normalized Ratio (INR) >1.5 × ULN
* MRI during the screening period showed heavy iron overload and is judged by the investigator to be unable to participate in the study.
* Patients with past/present history of cancer
* Known neurological disorders, psychological problems or mental illness, and is judged by the investigator to be unable to cooperate with the study procedures
* Known history of uncontrolled epileptic seizures and is judged by the investigator to be unfit to participate in this study
* Known history of other serious cardiovascular, pulmonary, renal diseases, digestive tract conditions, liver diseases and / or other conditions, etc., and are judged by the investigator to be intolerable or inappropriate for autologous hematopoietic stem cell mobilization, collection, and myeloablative conditioning and infusion
* Pregnant or lactating women

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events(AEs) as assessed by CTCAE v5.0 | From signing informed consent to 180 days post-CS-101 infusion
Occurrence of engraftment | within 42 days post-CS-101 infusion
  Subjects with engraftment is defined as neutrophil engrafted
Time to neutrophil and platelet engraftment | Days post-CS-101 infusion
  Time to neutrophil engraftment is defined as first day of 3 consecutive measurements of absolute neutrophil count≥0.5×10^9/L on three different days; Time to platelet engraftment is defined as first day of 3 consecutive measurements of absolute platelet count≥20×10^9/L on three different days and without platelet transfusion
Occurrence of transplant-related death | baseline to 100 days post-CS-101 infusion
Occurrence of all-cause death | From signing informed consent to 180 days post-CS-101 infusion
Occurrence of achieving transfusion reduction for at least 3 consecutive months | From 3 months post -CS-101 infusion to 3 months post -CS-101 infusion

SECONDARY OUTCOMES:
Occurrence of achieving transfusion independence for at least 3 consecutive months | From 3 months up to 180 days post-CS-101 infusion
Time to last red blood cell(RBC) transfusion | Days post-CS-101 infusion
Change in total hemoglobin(Hb) concentration over time | up to 180 days post-CS-101 infusion
Change in fetal hemoglobin(HbF) concentration over time | up to 180 days post-CS-101 infusion
Chimerism level in Peripheral blood and bone marrow | up to 180 days post-CS-101 infusion
  Proportion of alleles with intended genetic modification in peripheral blood leukocytes and bone marrow over time

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Zhai, M.D., Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No